CLINICAL TRIAL: NCT06723470
Title: Effect of Passive Smoking on Functional Capacity, Cognition and Academic Performance in Primary School Children
Status: Not yet recruiting | Type: Observational
Sponsor: Egyptian Chinese University (Other)
Responsible Party: Principal Investigator, Nourhan Abdelaleem, Assistant lecturer of Pediatric Physical Therapy, Egyptian Chinese University
Other Study IDs: P.T.REC/012/005358
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Smoke Exposure; Smokeless Tobacco
Keywords: Passive Smoking; Functional Capacity; Cognitive Abilities; Academic Performance; Children; Primary School; Physical Fitness
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Passive Smokers: This group includes children aged 6-11 years who are exposed to secondhand smoke at home. At least one parent or caregiver is a smoker, with a smoking history of no less than six years. The level of exposure is categorized as moderate to high based on the smoking index (number of cigarettes per day multiplied by years of smoking).
- Group 2: Non-Smokers: This group includes children aged 6-11 years who are not exposed to secondhand smoke at home or in other environments. Neither parent nor caregiver is a smoker, ensuring no passive smoke exposure.

SUMMARY:
This is an observational study that aims to understand the effects of passive smoking (secondhand smoke exposure) on children's health and development. The main question the study seeks to answer is:

How does exposure to secondhand smoke affect the physical fitness, cognitive abilities, and academic performance of primary school children?

The study will compare two groups of children aged 6-11 years: one group exposed to secondhand smoke at home (due to parents or caregivers who smoke) and another group not exposed to secondhand smoke. The children's physical capacity, cognitive skills, and school performance will be assessed through various tests.

The goal of the study is to provide valuable insights into how secondhand smoke may negatively impact children, helping families, schools, and healthcare providers understand the risks and promote healthier, smoke-free environments for children.

DETAILED DESCRIPTION:
This observational study aims to assess the effects of passive smoking on functional capacity, cognitive abilities, and academic performance in primary school children aged 6-11 years. The study will compare two groups: children exposed to secondhand smoke (passive smokers) and children not exposed (non-smokers).

Children in the passive smoking group have one or both parents who have been smoking for at least six years, with moderate to high levels of exposure based on a smoking index. These children will be compared with children in the non-smoking group who are not exposed to secondhand smoke at home or in other environments. The study will focus on three primary outcome areas:

* **Functional Capacity**: Measured by the 3-Minute Step Test to assess cardiorespiratory fitness and physical performance.
* **Cognitive Abilities**: Evaluated using the Wechsler Intelligence Scale for Children (WISC-V), which measures various cognitive functions, including verbal comprehension, working memory, and processing speed.
* **Academic Performance**: Assessed using the Academic Performance Rating Scale (APRS), which provides an evaluation of the child's academic success, attention, and classroom behavior.

This study will not involve any interventions, as it is observational in nature. Instead, it will collect data to identify differences in physical, cognitive, and academic outcomes based on passive smoking exposure. All data collection will occur at baseline, with the assessments conducted in a controlled, quiet environment to minimize distractions.

The sample will consist of 90 children (45 in each group), with participation based on inclusion and exclusion criteria. Children will be selected from primary schools in Cairo, Egypt, where parents have provided informed consent for participation. The study results will contribute valuable insights into the negative effects of secondhand smoke on children's health and development, which can guide health care providers, educators, and families in promoting smoke-free environments for children.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6-11 years, enrolled in primary school.
2. Both genders (male and female).
3. Healthy children with no musculoskeletal, visual, auditory, or cognitive impairments.
4. Children whose parents have been smoking for at least 6 years, with moderate to high smoking levels (based on the smoking index).
5. Children residing in a moderate socioeconomic status.
6. Children living in Cairo, Egypt.
7. Children who are able to follow simple commands and participate in assessments.

Exclusion Criteria:

1. Children with musculoskeletal problems, congenital deformities, visual or auditory defects, learning disabilities, or autism.
2. Children who are currently taking medications that affect alertness or cognitive function.
3. Children who are not exposed to secondhand smoke (non-smokers) but have parents who smoke at very low levels or do not meet the inclusion criteria for passive smoking exposure.
4. Children who are unable to cooperate or participate in the assessments.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consists of 90 primary school children aged 6-11 years, selected from various primary schools in Cairo, Egypt. These children are categorized into two groups: 45 children exposed to secondhand smoke (passive smokers) and 45 children not exposed to secondhand smoke (non-smokers). All children are healthy and without any cognitive, visual, or musculoskeletal impairments. The children in the passive smokers group have parents who have been smoking for at least 6 years with moderate to high levels of smoking exposure. The non-smokers group consists of children who are not exposed to secondhand smoke at home or in their environments. The children's participation is voluntary, with informed consent obtained from parents or guardians.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Impact of Passive Smoking on Functional Capacity in Primary School Children | At the start of the study (baseline).
  Functional capacity will be assessed using the 3-Minute Step Test (3MST). This test measures cardiorespiratory fitness by evaluating the total number of completed step cycles (up and down) within 3 minutes and the heart rate recovery one minute post-exercise. The reported outcomes will include:
  Number of steps completed (unit: step cycles). Heart rate recovery (unit: beats per minute). These outcomes will be analyzed separately. Higher heart rate recovery values indicate worse cardiorespiratory fitness, whereas more completed step cycles indicate better fitness.

SECONDARY OUTCOMES:
Impact of Passive Smoking on Cognitive Abilities in Primary School Children | At the start of the study (baseline).
  Cognitive abilities will be assessed using the Wechsler Intelligence Scale for Children (WISC-V). The WISC-V provides composite scores in five domains:
  Verbal Comprehension Index (VCI): range 50-150. Working Memory Index (WMI): range 50-150. Processing Speed Index (PSI): range 50-150. Fluid Reasoning Index (FRI): range 50-150. Full-Scale IQ (FSIQ): range 50-150. Higher scores indicate better cognitive functioning in each domain.
Impact of Passive Smoking on Academic Performance in Primary School Children | At the start of the study (baseline).
  Academic performance will be assessed using the Academic Performance Rating Scale (APRS). This scale includes 19 items, each rated on a 5-point Likert scale (1 = poor, 5 = excellent). The total score ranges from 19 to 95, with higher scores indicating better academic performance.

IPD SHARING:
Plan to Share IPD: Undecided